CLINICAL TRIAL: NCT06341764
Title: Neo-adjuvant Chemo and Immunotherapy with Durvalumab (MEDI4736) and Tremelimumab (MEDI1123) in the Pre-operAtive Treatment of Locally Advanced CholangIOcarciNoma: an Exploratory and Translational Study.
Brief Title: Neo-adjuvant Chemo and Immunotherapy in the Pre-operAtive Treatment of Locally Advanced CholangIOcarciNoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CITATION; 7/23 (Other: IRCCS I.N.T. "G. Pascale")
Record Dates: First submitted 2023-10-30; First posted 2024-04-02 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — durvalumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): Patient will receive four cycles of cisplatin (CDDP) 25 mg/mq i.v. and gemcitabine (GEM) 1000 mg/mq i.v. days 1 and 8 every 21 days, plus durvalumab 1120 mg day 1, followed (one week after the last dose of CDDP/GEM) by two administrations of durvalumab i.v. at 1500 mg once every 4 weeks and one administration of tremelimumab i.v. at 300 mg single dose. Premedication with antihistamines at standard doses can be applied.
  Interventions: Drug: Durvalumab 1120 mg; Drug: Durvalumab 1500 mg; Drug: Tremelimumab i.v. at 300 mg; Combination Product: Cisplatin (CDDP) 25 mg/mq i.v; Combination Product: Gemcitabine (GEM) 1000 mg/mq i.v.

INTERVENTIONS:
Drug: Durvalumab 1120 mg — Durvalumab 1120 mg day 1 i.v
Drug: Durvalumab 1500 mg — Durvalumab i.v. at 1500 mg once every 4 weeks
Drug: Tremelimumab i.v. at 300 mg — Single dose
Combination Product: Cisplatin (CDDP) 25 mg/mq i.v — Four cycles
Combination Product: Gemcitabine (GEM) 1000 mg/mq i.v. — Days 1 and 8 every 21 days

SUMMARY:
Neoadjuvant chemo- and immunotherapy ameliorate the recurrence rate of cholangiocarcinoma (CCA) at 12 months after surgery.

DETAILED DESCRIPTION:
Multicenter, single arm, phase II study

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* Histologically or pathologically confirmed CCA
* Age >18 years at time of study entry.
* Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Locally advanced disease (as assessed in multidisciplinary sessions).
* Life expectancy of at least 16 weeks.
* Body weight >30 kg
* Adequate normal organ and marrow function as defined below: Haemoglobin ≥9.0 g/dL
* Absolute neutrophil count (ANC ≥1.5 × 109 /L)
* Platelet count ≥100 × 109/L
* Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
* AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
* Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
* At least 1 lesion that qualifies as a RECIST 1.1 target lesion (TL) at baseline. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to randomization.
* No previous systemic or local treatments including radiation therapy, radiofrequency ablations, electro-chemotherapy.

Exclusion Criteria:

* Any previous participation in another clinical interventional study.
* Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, interstitial lung disease, etc.]). The following are exceptions to this criterion:

  1. Patients with vitiligo or alopecia
  2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  3. Any chronic skin condition that does not require systemic therapy
  4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  5. Patients with celiac disease controlled by diet alone
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, history of myocardial infarction within 12 months, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* History of bowel obstruction, refractory ascites, or bowel perforation due to advanced disease within the past 3 months from start of study treatment.
* Significant bleeding diathesis or coagulopathy. Serious, nonhealing wound, ulcer, or current healing fracture.
* History of another primary malignancy except for

  1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis
* Brain metastases or spinal cord compression. Patients with suspected brain metastases at screening should have an MRI (preferred) or CT each preferably with IV contrast of the brain prior to study entry.
* History of active primary immunodeficiency.
* Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion: Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection
* Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or180 days after the last dose of durvalumab and tremelimumab combination therapy.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of CCA | 24 months
  To determine whether neoadjuvant chemo- and immunotherapy decrease the recurrence rate of CCA at 12 months after surgery.

SECONDARY OUTCOMES:
Rate of R0 resections | 24 months
  Rate of R0 resections (number of resections with surgical margins free from cancer/total number of resections) as assessed by pathologic examination (R1: microscopic disease.
Radiologic responses | 24 months
  Radiologic responses evaluated through the RECIST v1.1 criteria.
Pathologic responses | 24 months
  Pathologic responses (number of surgically removed tumour specimens with absence of any residual viable neoplastic cells).
Toxicity assessed | 24 months
  Toxicity assessed by the NCI CTCAE v5.0
PFS | 24 months
  Progression free survival (PFS) measured from study enrolment to death
OS | 24 months
  Overall survival (OS) measured from study enrolment to death

OTHER OUTCOMES:
Exploratory objectives | 24 months
  Characterization of tumor microenvironment of primary CCAs and eventually resected metastases treated with neoadjuvant sequential chemo-immuno-therapy
Exploratory objectives | 24 months
  Depiction of mutational evolution of CCA through NGS (Next Generation Sequencing) gene analysis on primary tumor biopsies and matched metastases (FFPE tissues or liquid biopsies).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Ottaiano, Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (6):
- Italy (6):
  - Istituto Nazionale Tumori di Napoli - IRCCS - Fondazione G. Pascale, Napoli, Italia
  - Ospedale Cardarelli, Napoli, Napoli, Italia
  - Università di Napoli "Federico II", Napoli, Napoli, Italia
  - Ospedale san Camillo Forlanini/Spallanzani, Roma, Roma, Italia
  - Ospedale Mauriziano, Umberto I°, Torino, Italia
  - Università di Verona, Ospedale Borgoroma, Verona, Verona, Italia